CLINICAL TRIAL: NCT00113958
Title: Cinacalcet Open Label Study to Reach K/DOQI Levels
Brief Title: Cinacalcet Study to Reach Kidney Disease Outcomes Quality Initiative (K/DOQI) Levels
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20020389
Record Dates: First submitted 2005-06-10; First posted 2005-06-13 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: End Stage Renal Disease
Keywords: End Stage Renal Disease (ESRD); secondary hyperparathyroidism (SHPT); hemodialysis; biPTH; AMG 073, Amgen
MeSH Terms: conditions — Kidney Failure, Chronic; Hyperparathyroidism, Secondary | interventions — Cinacalcet

INTERVENTIONS:
Drug: Cinacalcet

SUMMARY:
The purpose of this study is to observe the effects of a treatment strategy that incorporates cinacalcet HCl into the management of secondary hyperparathyroidism (HPT) to K/DOQI recommended targets in subjects with end stage renal disease (ESRD) receiving hemodialysis, on bio-intact parathyroid hormone, corrected serum calcium, serum phosphorus, and calcium phosphorus product.

ELIGIBILITY:
Inclusion Criteria: - Men and women must agree to use highly effective contraceptive measures throughout the study - Prescribed hemodialysis for at least 3 months before study day 1 - Must be receiving IV vitamin D sterols during the 30 days before day

1 (greater than 2 µg of paricalcitol, greater than 1 µg of doxercalciferol, or greater than 0.5 µg of calcitriol per dialysis treatment) - The mean of 2 biPTH determinations obtained from the central laboratory must be greater than or equal to 80 pg/mL and less than or equal to 160 pg/mL - The mean 2 albumin corrected serum calcium determinations obtained from the central laboratory must be greater than or equal to 8.4 mg/dL - The mean of two Ca x P calculations, based on corrected serum calcium and serum phosphorus determinations obtained from the central laboratory must be greater than 55 mg²/dL Exclusion Criteria: - Have an unstable medical condition, defined as having been hospitalized, other than for dialysis vascular access revision, within 30 days before day 1, or otherwise unstable in the judgment of the investigator - Pregnant or nursing females - Parathyroidectomy in the 12 weeks before day 1 - Received, within 21 days before day 1 of the dose titration phase, therapy with medications that are predominantly metabolized by the enzyme CYP2D6 and have a narrow therapeutic index (e.g., flecainide, vinblastine, thioridazine and most tricyclic antidepressants). The antidepressant amitriptyline is permitted - Received, within 21 days before day 1, therapy with medications that are potent inhibitors (e.g., ketoconazole, itraconazole and erythromycin) or inducers (e.g., rifampin and St. John's Wort) of the enzyme CYP3A4. Phenytoin, phenobarbital and carbamazepine are also potent inducers of this enzyme. However, subjects on a stable dose of any of these anti-convulsants at baseline, with no evidence of seizure activity in the past 2 months may be eligible for the study - Experienced a myocardial infarction within 12 weeks prior to day 1 - Currently enrolled in, or have not yet completed at least 30 days since ending other investigational device or drug trials, or are receiving other investigational agents (experimental dialysis machines are acceptable) - Current gastrointestinal disorder that may be associated with impaired absorption of orally administered medications or an inability to swallow tablets - Participated in other studies with cinacalcet HCl - Disorder that would interfere with the understanding and giving of informed consent or compliance with protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Secondary hyperparathyroidism in people with kidney failure.

SECONDARY OUTCOMES:
Uncontrolled secondary hyperparathyroidism

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Chertow GM, Blumenthal S, Turner S, Roppolo M, Stern L, Chi EM, Reed J; CONTROL Investigators. Cinacalcet hydrochloride (Sensipar) in hemodialysis patients on active vitamin D derivatives with controlled PTH and elevated calcium x phosphate. Clin J Am Soc Nephrol. 2006 Mar;1(2):305-12. doi: 10.2215/CJN.00870805. Epub 2006 Jan 25. PMID 17699221
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com